CLINICAL TRIAL: NCT02741947
Title: Clinical and Pharmacokinetics Study to Evaluate the Therapeutic Equivalence and Bioequivalence of Levodopa Benserazide Generic Formulation (Teva Italia) Versus the Originator (Madopar®)
Brief Title: Levodopa Benserazide Generic Formulation Versus the Originator
Acronym: FARM9X59Y4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RP 13/12
Record Dates: First submitted 2016-03-31; First posted 2016-04-18 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2016-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Therapeutic Equivalence; Levodopa
MeSH Terms: conditions — Parkinson Disease | interventions — benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levodopa Benserazide Madopar (Active Comparator): Madopar 100+25mg and 200+50mg, tablet, tid e qid, for four weeks
  Interventions: Drug: Levodopa Benserazide Madopar
- Levodopa Benserazide Teva Italia (Experimental): Levodopa Benserazide Teva Italia100+25mg and 200+50mg, tablet, tid e qid, for four weeks
  Interventions: Drug: Levodopa Benserazide Teva Italia

INTERVENTIONS:
Drug: Levodopa Benserazide Madopar — Madopar 100+25mg and 200+50mg, tablet, tid e qid, for four weeks
  Arms: Levodopa Benserazide Madopar
Drug: Levodopa Benserazide Teva Italia — Levodopa benserazide Teva 100+25mg and 200+50mg, tablet, tid e qid, for four weeks
  Arms: Levodopa Benserazide Teva Italia

SUMMARY:
The trial was an experimental two-centers, randomized, double-blind, two-sequence, non-inferiority cross-over study.

Screened subjects already treated with Levodopa/Benserazide (LDB) (Madopar®) who agreed to participate in the study entered a 4 weeks period if not on stable regimen of Madopar® (run-in period). Following the run-in period, there were two maintenance periods of 4 weeks each, for a total duration of 8 weeks.

Patients were assigned randomly (1:1) by a computerized randomization system to one of two formulation sequences maintaining the dose stabilized during the run in:

* generic-originator
* originator-generic At the end of maintenance period 1, the patients in each formulation group underwent an overnight switch to the same dose of the alternative formulation. The dose was kept stable during the whole length of trial. Clinical evaluations were performed at the end of each period. The tablets were encapsulated to maintain the blindness.

A pharmacokinetic study with a fixed dose (100+25 mg) was performed in a sub-population of 14 subjects.

Population: out-patients with a diagnosis of idiopathic Parkinson's disease for at least 5 years, receiving L-dopa/benserazide.

The total duration of the trial was approximately 8 weeks for patient divided in two maintenance periods of 4 weeks each.

DETAILED DESCRIPTION:
The trial was an experimental two-centers, randomized, double-blind, two-sequence, non-inferiority cross-over study.

Population: out-patients with a diagnosis of idiopathic Parkinson's disease (PD) for at least 5 years, receiving Levodopa, were enrolled to participate into the study. The study was performed in hospital setting using the facilities of the clinical trial centre in both sites involved in the study. The patients were recruited within the patient population using the hospitals out-patients clinics. Recruitment timing lasted 18 months.

Screened subjects who agreed to participate in the study, taking Levodopa/Benserazide LDB (Madopar®) entered a 4 weeks period with stable regimen of Madopar® (run-in period). The formulations of levodopa admitted in the trial were: Madopar® 100+25; and 200+50 (1/2 or 1 tablet). Following the run-in period, there were two key phases of the study: two maintenance periods (4 weeks each), for a total duration of 8 weeks. Patients were assigned randomly (1:1) by a computerized randomization system to one of two formulation sequences maintaining the dose stabilized during the run in:

* generic-originator
* originator-generic At the end of maintenance period 1, the patients in each formulation group underwent an overnight switching to the same dose of the alternative formulation. The dose was kept stable during the whole length of trial. Clinical evaluations were performed at the end of each period (see flow chart enclosed). The tablets were encapsulated to maintain the blindness. A pharmacokinetic study with a fixed dose (100+25 mg) was performed in a sub-population of 14 subjects. The drugs was administered orally. In case of prolonged, not tolerable akinetic periods during the study, the patients could be rescued with an extra dose of levodopa. Any antiparkinsonian treatment modification or supplementation of antiparkinsonian drugs was not allowed during the study. Any other drug not specific for Parkinson's disease was evaluated by the investigators and allowed only if necessary and if not interfering with the study drugs.

The random allocation of patients to one of the two treatment groups was centrally managed by the coordinating centre, according to an automatically generated randomization list provided by the team responsible for the data collection monitoring and statistical analysis. An allocation ratio of 1:1 was assumed when generating the list. Patients eligible to enter the randomization procedure was sequentially assigned to the lowest randomization sequence number not yet assigned to any study subject. For each randomization number, a sealed envelope containing the randomization code was prepared by the team that generated the randomization list. Unblinding was permitted only if strictly necessary. In case it was essential to know the treatment assigned to a patient due to serious unexpected adverse events, the envelope containing the patient's randomization code could be open. In such cases, a detailed report on the timing, the causes and the patient's randomization number would have been issued by the person responsible for the trial and archived by the coordinating centre.

Mechanical blinding (encapsulation) was used to ensure the double-blind nature of the study. Because the patients enrolled in the trial received levodopa/benserazide in different doses, over-encapsulation of tablets permitted blinding of most oral dosage forms: ½ tablet, several small tablets, capsules of different sizes or colors. Each capsule was then be placed in a narrow opaque tube and identified as "Treatment 1" and "Treatment 2" before administration to the patient. The patient, the investigator, Medical Monitor and Clinical Monitor remained blinded, whereas the site pharmacist and a nurse who administered study medication were not blind throughout this part of the study.

No interim analysis was planned for this protocol. Amendments: no amendments were presented during the study.

ELIGIBILITY:
Inclusion Criteria

Out-patients with a diagnosis of idiopathic Parkinson's disease for at least 5 years, receiving L-dopa/benserazide, were enrolled to participate into the study. The patients were recruited within the patient population using the hospitals out-patients clinics.

* Subject must be ≥30 and ≤75 years of age, of either sex and of any race.
* Diagnosis of Parkinson's disease
* Subjects in Hoehn and Yahr stages 2 to 4.
* Subject must have good response to levodopa (≥30% improvement in the UPDRS score).
* Subject must have been on a stable regimen of L-dopa for at least 4 month before Screening.
* A female subject must be postmenopausal, or sterile or use a medically accepted method of contraception.

Fragile population was included in the trial (Elderly 65-74 years and over 75 years).

Exclusion Criteria

* Atypical Parkinsonism
* Subjects with very severe motor fluctuations and/or dyskinesias.
* Significant internal-medicine or psychiatric diseases.
* Subject's clinical laboratory tests outside the normal ranges.
* History of previous rhabdomyolysis
* Subjects in therapy with Catechol-O-methyltransferase-inhibitor.
* Subjects who participated in any other clinical trial in the 4 months before the screening.
* Any subject who is pregnant or breastfeeding.
* Subjects demented or not able to give informed consent to trial

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in bioequivalence in the total Area Under the Curve (AUC-t) between the generic levodopa/benserazide and the originator. | end of maintenance period 1 and maintenance period 2 (each period of 4 weeks)
  AUC-t: area under the curve within first and last observed point
Change in therapeutic equivalence measured with the Unified Parkinson's Disease rating scale part III between the generic levodopa/benserazide and the originator. | end of maintenance period 1 and maintenance period 2 (each period of 4 weeks)
  A difference of -3 points on the UPDRS motor score be the margin for non-inferiority

SECONDARY OUTCOMES:
Change in Patient Clinical Global Impression - Global Improvement scale between the generic levodopa/benserazide and the originator. | end of maintenance period 1 and maintenance period 2 (each period of 4 weeks)
Change in bioequivalence in minimum concentration (Cmin) between the generic levodopa/benserazide and the originator. | end of maintenance period 1 and maintenance period 2 (each period of 4 weeks)
Change in bioequivalence in time to maximum concentration (Tmax) after the last dose between the generic levodopa/benserazide and the originator. | end of maintenance period 1 and maintenance period 2 (each period of 4 weeks)
Change in bioequivalence in the half life (t 1/2) after the last dose between the generic levodopa/benserazide and the originator. | end of maintenance period 1 and maintenance period 2 (each period of 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: FABRIZIO STOCCHI, PROFESSOR, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Irccs San Raffaele Pisana, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stocchi F, Jenner P, Obeso JA. When do levodopa motor fluctuations first appear in Parkinson's disease? Eur Neurol. 2010;63(5):257-66. doi: 10.1159/000300647. Epub 2010 Mar 24. PMID 20332641
- [Result] Olanow CW, Agid Y, Mizuno Y, Albanese A, Bonuccelli U, Damier P, De Yebenes J, Gershanik O, Guttman M, Grandas F, Hallett M, Hornykiewicz O, Jenner P, Katzenschlager R, Langston WJ, LeWitt P, Melamed E, Mena MA, Michel PP, Mytilineou C, Obeso JA, Poewe W, Quinn N, Raisman-Vozari R, Rajput AH, Rascol O, Sampaio C, Stocchi F. Levodopa in the treatment of Parkinson's disease: current controversies. Mov Disord. 2004 Sep;19(9):997-1005. doi: 10.1002/mds.20243. PMID 15372588
- [Result] Stocchi F. The levodopa wearing-off phenomenon in Parkinson's disease: pharmacokinetic considerations. Expert Opin Pharmacother. 2006 Jul;7(10):1399-407. doi: 10.1517/14656566.7.10.1399. PMID 16805724